CLINICAL TRIAL: NCT04467034
Title: A Randomized Controlled Trial to Evaluate The Stanford Tobacco Prevention Toolkit
Brief Title: Evaluation of The Stanford Tobacco Prevention Toolkit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Schools were unable to participate due the COVID-19 pandemic, which shifted educational priorities and therefore impeded school-based recruiting efforts. No participants were enrolled.
Sponsor: Stanford University (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Principal Investigator, Bonnie Halpern-Felsher, Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 54817
Record Dates: First submitted 2020-05-21; First posted 2020-07-10 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Behavior, Health; Behavior, Smoking
Keywords: children; young adults; tobacco; education; health; smoking; prevention
MeSH Terms: conditions — Health Behavior; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receives Stanford tobacco education curriculum (Experimental): Stanford Tobacco Prevention Toolkit is administered.
  Interventions: Behavioral: Stanford Tobacco Prevention Toolkit curriculum
- Does not receive Stanford tobacco education curriculum (No Intervention): Receives another curriculum or no tobacco education.

INTERVENTIONS:
Behavioral: Stanford Tobacco Prevention Toolkit curriculum — Stanford Toolkit curriculum delivered as a 5-session course in a school classroom setting.
  Arms: Receives Stanford tobacco education curriculum

SUMMARY:
The Stanford Tobacco Prevention Toolkit is a free online curriculum developed for use by educators and health professionals in providing tobacco-specific prevention education to middle and high school students. The aims of this study are to determine: (1) whether the Curriculum is effective in changing middle and high school students' resistance to using tobacco as well as knowledge of, attitudes towards, and intentions to use different tobacco products; and (2) whether the Curriculum is effective in changing middle and high school students' actual use of tobacco in the short-term.

ELIGIBILITY:
Inclusion Criteria:

* Middle school and high school students

Exclusion Criteria:

* Non English-speakers

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in resistance to use of tobacco products scaled score as measured by investigator-originated survey | Change from baseline to follow-up at approximately 40 weeks post-baseline
  This survey measures change in resistance to use of tobacco products with questions related to the participant's intention to use tobacco.

SECONDARY OUTCOMES:
Change in skills for refusal of tobacco products scaled score as measured by investigator-originated survey | Change from baseline to follow-up at approximately 40 weeks post-baseline
  This survey measures change in skills to refuse tobacco use with questions related to the participant's susceptibility to tobacco use, self-efficacy and self-confidence.
Change in knowledge of tobacco products scaled score as measured by investigator-originated survey | Change from baseline to follow-up at approximately 40 weeks post-baseline
  This survey measures knowledge of tobacco products with questions related to the participant's knowledge of ingredients, of nicotine levels, of potential health outcomes.
This survey measures use of tobacco products with questions related to the participant's ever tobacco use, past 30-day tobacco use, and past 7-day tobacco use. | Change from baseline to follow-up at approximately 40 weeks post-baseline
  Investigator-originated survey survey measures (questions) assess ever tobacco use, past 30-day tobacco use, past 7-day tobacco use This outcome measure assesses tobacco products use.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie L Halpern-Felsher, Principal Investigator — Stanford School of Medicine, Department of Pediatrics; Michael Baiocchi, Principal Investigator — Stanford School of Medicine, Department of Epidemiology and Population Health
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Stanford Tobacco Prevention Toolkit — https://med.stanford.edu/tobaccopreventiontoolkit.html